CLINICAL TRIAL: NCT06855888
Title: Comparison of Three-sided and Single-sided Mattress Pancreaticojejunostomy in Pancreatoduodenectomy -Randomized Controlled Trial-
Brief Title: Comparison of Three-sided and Single-sided Mattress Pancreaticojejunostomy in Pancreatoduodenectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tokai University (Other)
Responsible Party: Principal Investigator, Ken-ichi Okada, Professor, Tokai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24R128; UMIN000056623 (Other: University Hospital Medical Information Network Clinical Trials Registry (UMIN))
Record Dates: First submitted 2025-02-21; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pancreatic Fistula Post-pancreatoduodenectomy
Keywords: mattress suture; pancreaticojejunostomy; pancreatoduodenectomy; postoperative pancreatic fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Once PD is performed, there is no difference in postoperative radiographic findings between the two surgical approaches, so it should not affect the radiologist's assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Modified Blumgart suture method (conventional treatment group) (Placebo Comparator)
  Interventions: Procedure: Modified Blumgart suture method
- Group B: Three-sided mattress suture (test treatment group) (Active Comparator)
  Interventions: Procedure: Three-sided mattress suture

INTERVENTIONS:
Procedure: Modified Blumgart suture method — During pancreaticoduodenectomy, the modified Blumgart suture method is used for pancreaticojejunostomy. For anastomosis, 5-0PDS is used for pancreatic duct mucosal anastomosis, and 3-0 or 4-0 monofilament non-absorbable suture is used for pancreaticojejunal mattress anastomosis.
  Arms: Group A: Modified Blumgart suture method (conventional treatment group)
Procedure: Three-sided mattress suture — At the time of pancreaticoduodenectomy, the three-sided mattress suture is used as the pancreaticojejunostomy method. In addition to the conventional Blumgart modified suture, the three-sided mattress suture method adds a mattress anastomosis with 3-0 or 4-0 monofilament non-absorbable suture to the cranial and caudal sides of the pancreaticojejunostomy site.
  Arms: Group B: Three-sided mattress suture (test treatment group)

SUMMARY:
In pancreaticojejunostomy following pancreaticoduodenectomy for soft pancreas, a randomized controlled trial will be conducted to compare a patient group using the conventional Blumgart modified technique and a patient group in which mattress sutures are added to the cranial and caudal sides of the pancreaticojejunostomy after the Blumgart modified technique (three-sided mattress suture technique), and to evaluate the safety and usefulness of the three-sided mattress suture technique by comparing the incidence of pancreatic fistula (ISGPF grade B or C).

DETAILED DESCRIPTION:
Pancreatoduodenectomy (PD) is one of the most difficult and invasive surgeries, with a 30-50% complication rate even at high volume centers. In particular, if a postoperative pancreatic fistula (POPF), a failure of the pancreaticojejunostomy (PJ) suture, occurs, pancreatic juice containing powerful digestive enzymes leaks into the abdominal cavity, which can develop into serious complications such as intraperitoneal abscesses and postpancreatectomy hemorrhage. To reduce the incidence of POPF post-PD, many clinical studies have been reported on PJ methods. Currently, the original/modified Blumgart method is widely used as an anastomosis technique with relatively good results, but the incidence of International Study Group for Pancreatic Surgery (ISGPS) criteria grade B/C is still around 10-20%. In particular, the incidence of POPF grade B/C in normal soft pancreases with preserved pancreatic function is high at approximately 20-40%, and it is known to be a higher risk than the atrophied, sclerosing pancreas after pancreatitis (incidence rate of approximately 0-10%), and there is still room for improvement in the PJ technique. Therefore, the current clinical problem to be solved in PD is "PJ for the soft pancreas," and reducing the incidence of POPF is thought to be extremely beneficial for patients.

In recent years, it has been reported that the incidence of pseudoaneurysm increases significantly when POPF is found on the superior side of the PJ, and that the incidence of deep surgical site infection increases when POPF occurs on the inferior side of the anastomosis. In the Blumgart method, ventral and dorsal sides of the pancreatic stump are covered by the jejunal wall, but a weak point remains where the jejunal wall does not completely cover the superior and inferior sides of the PJ anastomosis. Therefore, the investigators created a three-sided mattress suture method to eliminate weak gaps by adding mattress sutures between the pancreas and jejunum on the superior and inferior sides of the PJ anastomosis to reduce the incidence of grades B/C POPF.

Prior to this study, the investigators conducted a pilot study in which a three-sided mattress suture was performed for PJ following pylorus-resecting PD in 10 consecutive patients with soft pancreases, and no case of POPF ISGPF grade B/C was observed (incidence rate 0%). The Three-sided mattress method is original, and no randomized controlled trial has proven that this novel method contributes to improving the incidence of POPF post-PD. In this study, the investigators conducted a randomized controlled phase II trial comparing the three-sided mattress suture method with the conventional modified Blumgart suture method, with the aim of proving the effectiveness of this original suture method by examining the incidence of POPF grade B/C. If the usefulness of the three-sided mattress suture method is proven in this study, it is expected to have a major impact as a safer PJ method in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for pancreaticoduodenectomy who have been determined to have a soft pancreas.
2. Preoperative CT images show that the pancreatic duct diameter at the planned site of pancreatic resection is 5mm or less.
3. ECOG Performance Status (PS) is 0-1.
4. Age 18 years or older.
5. Function of major organs (bone marrow, heart, liver, kidneys, lungs, etc.) is maintained.
6. Patients have sufficient judgment to understand the content of the research, and written consent has been obtained from the individual.

Exclusion Criteria:

1. Patients with severe ischemic heart disease
2. Patients with liver cirrhosis or active hepatitis
3. Patients with respiratory distress requiring oxygen due to interstitial pneumonia or pulmonary fibrosis
4. Patients undergoing dialysis due to chronic renal failure
5. Patients requiring combined resection of surrounding organs
6. Patients requiring arterial reconstruction of the superior mesenteric artery, common hepatic artery, celiac artery, etc.
7. Patients with active duplicate cancers that may affect adverse events or overall survival
8. Patients taking oral steroids for a long period that may affect adverse events
9. Patients with insufficient decision-making ability
10. Other subjects deemed inappropriate by the principal investigator or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula ISGPF grade B or C | Up to 90 days after surgery

SECONDARY OUTCOMES:
Incidence of postoperative complications, incidence of remnant pancreatitis | Up to 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tokai University, Isehara-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Undecided